CLINICAL TRIAL: NCT07084246
Title: A Multi-center, Prospective, Non-intervention, Observational Study to Evaluate the Effectiveness and Safety of the Rozetel Tablet in Patients Who Had Undergone Percutaneous Coronary Intervention(PCI)
Brief Title: Evaluation of the Effectiveness and Safety of Rozetel Tablet in Patients After PCI: A Multi-Center Observational Study
Status: Active, not recruiting | Type: Observational
Sponsor: GC Biopharma Corp (Industry)
Responsible Party: Sponsor
Other Study IDs: GC7007_PCI_P4o01
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Hypertension, Dyslipidemia
MeSH Terms: conditions — Hypertension; Dyslipidemias

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of the investigational drug on blood pressure and LDL cholesterol control during the observation period in patients who have undergone percutaneous coronary intervention (PCI) in actual clinical practice.

DETAILED DESCRIPTION:
This study is a multicenter, prospective, non-interventional observational study aimed at observing the efficacy and safety of the investigational product, a combination of telmisartan, rosuvastatin, and ezetimibe, in patients who have undergone percutaneous coronary intervention (PCI) for the control of blood pressure and lipid levels.

In actual clinical practice, patients aged 19 years and older who have undergone PCI and are receiving antihypertensive and dyslipidemia-related medications based on approved indications will be assessed for eligibility after receiving an explanation of the study and providing written consent, as determined by the investigator's judgment regarding the need for the investigational product.

Eligible participants according to the inclusion/exclusion criteria will receive the investigational product based on the approved indications (efficacy, dosage, precautions, etc.) after registration. Follow-up visits will be conducted at 24 weeks and 48 weeks (each ± 4 weeks) post-treatment to evaluate efficacy and safety.

All treatments, including drug administration and laboratory tests performed after the administration of the investigational product, will be conducted according to the investigator's medical judgment, independent of the participant's involvement in the study, and information to be collected in this observational study will continue for up to 48 weeks (± 4 weeks).

ELIGIBILITY:
Inclusion Criteria:

* 1. Adults aged 19 years and older, both male and female. 2. Patients who have undergone percutaneous coronary intervention (PCI) and are receiving antihypertensive and dyslipidemia-related medications.

  3. Individuals who require the administration of the investigational product based on the investigator's medical judgment in accordance with approved indications.

  4. Individuals who can understand the information provided to them and are able to voluntarily sign the informed consent form.

Exclusion Criteria:

* 1. Individuals who fall under the contraindications for administration according to the approved indications of the investigational product.

  2. Individuals who have a history of receiving the investigational product prior to participation in this study.

  3. Individuals whom the investigator deems unsuitable for participation in this observational study for any other reason.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A patient population with a history of undergoing PCI
Sampling Method: Probability Sample
Enrollment: 1563 (Actual)
Dates: Start 2023-06-07 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The proportion of participants who meet the treatment goals for BP and LDL-C | From enrollment to the end of treatment at 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- GC Biopharma, Yŏngin, South Korea

IPD SHARING:
Plan to Share IPD: Undecided